CLINICAL TRIAL: NCT00005542
Title: Sarcoid Genetic Analysis (SAGA)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5084; U01HL060263 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-10

CONDITIONS: Lung Diseases; Sarcoidosis
MeSH Terms: conditions — Lung Diseases; Sarcoidosis

SUMMARY:
To identify sarcoidosis susceptibility genes and to determine how these genes and environmental risk factors interact to cause sarcoidosis.

DETAILED DESCRIPTION:
BACKGROUND:

Sarcoidosis is a rare systemic granulomatous disease that mainly affects young to middle aged adults, and more severely affects African Americans than Caucasians. The etiology of sarcoidosis is not yet known, and epidemiological studies have only identified general risk factors including age, sex, race, and family history. Sarcoidosis may also be influenced by environmental factors, although the particular environmental agents have not yet been clearly defined. While previous studies have provided evidence for familial clustering, little is known about the genes that influence predisposition to sarcoidosis.

DESIGN NARRATIVE:

This is a multicenter consortium genetic epidemiology study. The investigators will accomplish their goal by organizing a 10-site multi-center consortium to recruit an adequate sample of sarcoidosis families for analysis. They plan to use the affected sibling pair linkage analysis to scan the genome for linked chromosomal regions, transmission disequilibrium testing to evaluate candidate genes in those regions with evidence for linkage, and an environmental questionnaire to collect data to test for possible interactions of susceptibility genes with exogenous risk factors. Genotyping and analysis of data are scheduled to begin in July, 2001 with completion of all analysis by April, 2004.

The study consists of a Clinical Core, a Data Coordinating Core, and a Genetics Core with a DNA Processing Center and a Genotyping Center. Eight of the ten clinical centers comprising the Clinical Core are members of the ACCESS, A Case Control Etiology of Sarcoidosis Study.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-05; Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Iannuzzi — Henry Ford Hospital

REFERENCES:
- [Background] Maliarik MJ, Chen KM, Sheffer RG, Rybicki BA, Major ML, Popovich J Jr, Iannuzzi MC. The natural resistance-associated macrophage protein gene in African Americans with sarcoidosis. Am J Respir Cell Mol Biol. 2000 Jun;22(6):672-5. doi: 10.1165/ajrcmb.22.6.3745. PMID 10837363
- [Background] Rybicki BA, Walewski JL, Maliarik MJ, Kian H, Iannuzzi MC; ACCESS Research Group. The BTNL2 gene and sarcoidosis susceptibility in African Americans and Whites. Am J Hum Genet. 2005 Sep;77(3):491-9. doi: 10.1086/444435. Epub 2005 Jul 20. PMID 16080124
- [Background] Rybicki BA, Hirst K, Iyengar SK, Barnard JG, Judson MA, Rose CS, Donohue JF, Kavuru MS, Rabin DL, Rossman MD, Baughman RP, Elston RC, Maliarik MJ, Moller DR, Newman LS, Teirstein AS, Iannuzzi MC. A sarcoidosis genetic linkage consortium: the sarcoidosis genetic analysis (SAGA) study. Sarcoidosis Vasc Diffuse Lung Dis. 2005 Jun;22(2):115-22. PMID 16053026